CLINICAL TRIAL: NCT05126433
Title: EMERGE-201: A Phase 2, Multicenter, Open-label Study of Lurbinectedin Efficacy and Safety in Participants With Advanced or Metastatic Solid Tumors
Brief Title: Lurbinectedin Monotherapy in Participants With Advanced or Metastatic Solid Tumors
Acronym: JAZZ EMERGE201
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Termination of this study was a business decision made during portfolio review.
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: Jazz Pharmaceuticals Ireland Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JZP712-201
Record Dates: First submitted 2021-11-08; First posted 2021-11-19 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor; Urothelial Cancer; Poorly Differentiated Neuroendocrine Carcinomas; Homologous Recombination Deficient-Positive Malignancies Agnostic
Keywords: Lurbinectedin; Monotherapy; Urothelial cancer; Poorly differentiated neuroendocrine carcinomas; Homologous recombination deficient-positive malignancies agnostic
MeSH Terms: conditions — Neoplasm Metastasis | interventions — PM 01183

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Urothelial Cancer Cohort (Experimental): Participants with advanced (metastatic and/or unresectable) urothelial carcinoma who have progressed on platinum-containing regimen (prior therapies may include but are not limited to immune checkpoint inhibitor, enformumab vendotin, or sacituzumab govitecan) will receive Lurbinectedin 3.2 mg/m^2 intravenous (IV) on Day 1 of every 3 weeks (Q3W) cycle until confirmed disease progression, withdrawal of participant consent, participant lost to follow-up, unacceptable toxicity, or the study or individual cohort may be terminated by the sponsor for lack of efficacy signal or any other reason.
  Interventions: Drug: Lurbinectedin
- Poorly Differentiated Neuroendocrine Carcinomas Cohort (Experimental): Participants with advanced (metastatic and/or unresectable) poorly differentiated neuroendocrine carcinomas who received at least 1 prior line of therapy will receive Lurbinectedin 3.2 mg/m^2 intravenous (IV) on Day 1 of every 3 weeks (Q3W) cycle until confirmed disease progression, withdrawal of participant consent, participant lost to follow-up, unacceptable toxicity, or the study or individual cohort may be terminated by the sponsor for lack of efficacy signal or any other reason.
  Interventions: Drug: Lurbinectedin
- Homologous Recombination Deficient-Positive Malignancies Agnostic Cohort (Experimental): Participants with advanced (metastatic and/or unresectable) endometrial, biliary tract, urothelial, breast (TNBC or HR+HER2- breast cancer), pancreas, gastric, or esophageal solid tumors with preidentified germline and/or somatic pathogenic mutation and received at least 1 prior line of therapy will receive Lurbinectedin 3.2 mg/m^2 intravenous (IV) on Day 1 of every 3 weeks (Q3W) cycle until confirmed disease progression, withdrawal of participant consent, participant lost to follow-up, unacceptable toxicity, or the study or individual cohort may be terminated by the sponsor for lack of efficacy signal or any other reason.
  Interventions: Drug: Lurbinectedin

INTERVENTIONS:
Drug: Lurbinectedin — Lurbinectedin 3.2 mg/m^2 intravenous (IV) every 3 weeks (Q3W)

SUMMARY:
This is an open-label, multicenter, phase 2 study of lurbinectedin monotherapy in participants with advanced (metastatic and/or unresectable) solid tumors.

DETAILED DESCRIPTION:
This phase 2, multicenter, open-label study is designed to assess the safety and efficacy of lurbinectedin monotherapy in 3 cohorts of participants with high-unmet medical need: advanced (metastatic and/or unresectable) urothelial cancer (UC), poorly differentiated neuroendocrine carcinomas (PD-NEC), and a homologous recombination deficient-positive malignancies agnostic cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. ≥ 18 years of age
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Adequate organ and bone marrow function
5. Has measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
6. Have advanced (metastatic/unresectable) cancers in one of the following:

   1. Histologically or cytologically confirmed urothelial cancer
   2. Histologically or cytologically confirmed poorly differentiated neuroendocrine carcinoma
   3. Histologically or cytologically confirmed homologous recombination deficient-positive malignancies agnostic, which may include endometrial, biliary tract, urothelial, breast (TNBC or HR+HER2- breast cancer), pancreas, gastric, or esophageal solid tumors with preidentified germline and/or somatic pathogenic mutation
7. Adequate contraceptive precautions

Exclusion Criteria:

1. Known symptomatic central nervous system (CNS) metastasis requiring steroids
2. History of prior malignancy within 2 years of enrollment
3. Clinically significant cardiovascular disease
4. Active infection requiring systemic therapy
5. Significant non-neoplastic liver disease
6. Prior treatment with trabectedin or lurbinectedin
7. Treatment with an investigational agent within 4 weeks of enrollment
8. Received live vaccine with 4 weeks of first dose
9. Prior allogeneic bone marrow or solid organ transplant
10. Positive hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening
11. Positive human immunodeficiency virus (HIV) infection at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Stanford Cancer Center, Stanford, California
  - Eastern Connecticut Hematology and Oncology, Norwich, Connecticut
  - Florida Cancer Specialists, Fort Myers, Florida
  - Sarah Cannon, Florida Cancer Specialist, St. Petersburg, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Pikeville Medical Center, Pikeville, Kentucky
  - Dana Farber, Boston, Massachusetts
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Sarah Cannon, Zangmeister Cancer Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center Investigational Drug Service, Pittsburgh, Pennsylvania
  - Bon Secours Hematology and Oncology, Greenville, South Carolina
  - Sarah Cannon, Tennesse Oncology, Nashville, Tennessee
  - MD Anderson, Houston, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes
In accordance with ICMJE requirements, Jazz Pharmaceuticals may provide qualified external researchers access to individual participant data (IPD) and clinical trial data that underlie the results of this trial upon request. Qualified researchers can submit a request on https://www.jazzpharma.com/science/clinical-trial-data-sharing/ as outlined. Jazz Pharmaceuticals reserves the right not to consider a request. For inquiries about Jazz's data sharing policy contact clinicaldatasharing@jazzpharma.com.
URL: https://www.jazzpharma.com/science/clinical-trial-data-sharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 47 participants who met all eligibility criteria were enrolled and received treatment were included
Groups:
- Urothelial Cancer (UC) Cohort: Participants with advanced (metastatic and/or unresectable) urothelial carcinoma who have progressed on platinum-containing regimen (prior therapies may include but are not limited to immune checkpoint inhibitor, enformumab vendotin, or sacituzumab govitecan) will receive Lurbinectedin 3.2 mg/m^2 intravenous (IV) on Day 1 of every 3 weeks (Q3W) cycle until confirmed disease progression, withdrawal of participant consent, participant lost to follow-up, unacceptable toxicity, or the study or individual cohort may be terminated by the sponsor for lack of efficacy signal or any other reason.
- Poorly Differentiated Neuroendocrine Carcinomas (PD-NEC) Cohort: Participants with advanced (metastatic and/or unresectable) poorly differentiated neuroendocrine carcinomas who received at least 1 prior line of therapy will receive Lurbinectedin 3.2 mg/m^2 intravenous (IV) on Day 1 of every 3 weeks (Q3W) cycle until confirmed disease progression, withdrawal of participant consent, participant lost to follow-up, unacceptable toxicity, or the study or individual cohort may be terminated by the sponsor for lack of efficacy signal or any other reason.
- Homologous Recombination Deficient-Positive Malignancies Agnostic (HRD) Cohort: Participants with advanced (metastatic and/or unresectable) endometrial, biliary tract, urothelial, breast (TNBC or HR+HER2- breast cancer), pancreas, gastric, or esophageal solid tumors with preidentified germline and/or somatic pathogenic mutation and received at least 1 prior line of therapy will receive Lurbinectedin 3.2 mg/m^2 intravenous (IV) on Day 1 of every 3 weeks (Q3W) cycle until confirmed disease progression, withdrawal of participant consent, participant lost to follow-up, unacceptable toxicity, or the study or individual cohort may be terminated by the sponsor for lack of efficacy signal or any other reason.
Period: Overall Study
Arm/Group | Urothelial Cancer (UC) Cohort | Poorly Differentiated Neuroendocrine Carcinomas (PD-NEC) Cohort | Homologous Recombination Deficient-Positive Malignancies Agnostic (HRD) Cohort
Started | 15 | 12 | 20
Completed | 0 | 0 | 0
Not Completed | 15 | 12 | 20
Not completed — Withdrawal by Subject | 3 | 0 | 4
Not completed — Death | 9 | 3 | 5
Not completed — Study Terminated by sponsor | 0 | 1 | 2
Not completed — Progressive Disease | 1 | 4 | 3
Not completed — Sponsor decision- no further OS follow up required | 2 | 4 | 6

BASELINE CHARACTERISTICS:
Population: The baseline demographic characteristics were assessed in the Safety Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Urothelial Cancer (UC) Cohort | Poorly Differentiated Neuroendocrine Carcinomas (PD-NEC) Cohort | Homologous Recombination Deficient-Positive Malignancies Agnostic (HRD) Cohort | Total
Number analyzed (Participants) | 15 | 12 | 20 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 11 | 23
  >=65 years | 8 | 7 | 9 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 12 | 18
  Male | 14 | 7 | 8 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 3
  Not Hispanic or Latino | 15 | 9 | 18 | 42
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 4
  White | 11 | 8 | 17 | 36
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Investigator-Assessed Objective Response Rate (ORR) According to Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1
Description: The ORR is defined as the proportion of participants whose best overall response (BOR) is investigator-assessed confirmed complete response (CR) or partial response (PR) using the RECIST v1.1 criteria. BOR is defined as the best response recorded between the date of first dose and the date of objectively documented progression per RECIST v1.1, or the date of subsequent anticancer therapy, death due to any cause, loss to follow-up, or study discontinuation, whichever occurs first.
Time Frame: Baseline to disease progression or death, up to 36 weeks.
Population: Assessed in participants with available data in the Efficacy Analysis Set. To be included in the Efficacy Analysis Set, participant must have a measurable disease at baseline and one of the following: a) at least 1 post-baseline tumor assessment, b) clinical progression, or c) death. One participant in the HRD Cohort was not included in the Efficacy Analysis Set due to not meeting the criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Urothelial Cancer (UC) Cohort | Poorly Differentiated Neuroendocrine Carcinomas (PD-NEC) Cohort | Homologous Recombination Deficient-Positive Malignancies Agnostic (HRD) Cohort
Number analyzed (Participants) | 15 | 12 | 19
Participants | 0 | 2 | 1

2. Secondary Outcome: Investigator-Assessed Progression Free Survival (PFS) as Assessed Per Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1
Description: PFS is defined as the time from the first dosing date to the date of first documented disease progression or death due to any cause, whichever occurs first.
Time Frame: Baseline to disease progression or death, up to 36 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Urothelial Cancer (UC) Cohort | Poorly Differentiated Neuroendocrine Carcinomas (PD-NEC) Cohort | Homologous Recombination Deficient-Positive Malignancies Agnostic (HRD) Cohort
Number analyzed (Participants) | 15 | 12 | 19
months | 1.46 [0.89 to 3.32] | 2.07 [1.18 to 2.89] | 1.38 [1.35 to 2.79]

3. Secondary Outcome: Investigator-Assessed Time-To-Response (TTR) as Assessed Per Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1
Description: TTR is defined as the time from the first dosing date to the date of the first confirmed response (complete response [CR] or partial response [PR]), as assessed by the investigators.
Time Frame: Baseline to disease progression or death, up to 36 weeks
Population: Only study treatment responders were included in the data set. There were no responders in the UC cohort, 2 responders in the PD-NEC cohort and 1 in the HRD cohort.
Measure: Median (Full Range); unit: months
Arm/Group | Urothelial Cancer (UC) Cohort | Poorly Differentiated Neuroendocrine Carcinomas (PD-NEC) Cohort | Homologous Recombination Deficient-Positive Malignancies Agnostic (HRD) Cohort
Number analyzed (Participants) | 0 | 2 | 1
months |  | 2.76 [2.7 to 2.8] | 1.31

4. Secondary Outcome: Investigator-Assessed Duration of Response (DOR) as Assessed Per Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1
Description: DOR is defined as the time from the first confirmed response (complete response [CR] or partial response [PR]) to the date of the first documented tumor progression as determined using RECIST v1.1 criteria or death due to any cause, whichever occurs first
Time Frame: Baseline to disease progression or death, up to 36 weeks
Population: as for outcome 3
Measure: Median (Full Range); unit: months
Arm/Group | Urothelial Cancer (UC) Cohort | Poorly Differentiated Neuroendocrine Carcinomas (PD-NEC) Cohort | Homologous Recombination Deficient-Positive Malignancies Agnostic (HRD) Cohort
Number analyzed (Participants) | 0 | 2 | 1
months |  | 5.67 [2.8 to 8.6] | 2.79

5. Secondary Outcome: Investigator-assessed Disease Control Rate (DCR) as Assessed Per Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1
Description: DCR is defined as the proportion of participants whose best overall response (BOR) is confirmed complete response (CR), or partial response (PR), or stable disease (SD) using the RECIST v1.1 criteria.
Time Frame: Baseline to disease progression or death, up to 36 weeks.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Urothelial Cancer (UC) Cohort | Poorly Differentiated Neuroendocrine Carcinomas (PD-NEC) Cohort | Homologous Recombination Deficient-Positive Malignancies Agnostic (HRD) Cohort
Number analyzed (Participants) | 15 | 12 | 19
Participants | 4 | 5 | 7

6. Secondary Outcome: Overall Survival (OS) in Participants Treated With Lurbinectedin
Description: OS is defined as the time from the first dosing date to the date of death from any cause. A participant who has not died will be censored at the last known alive date
Time Frame: Baseline and every 3 months, up to 16 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Urothelial Cancer (UC) Cohort | Poorly Differentiated Neuroendocrine Carcinomas (PD-NEC) Cohort | Homologous Recombination Deficient-Positive Malignancies Agnostic (HRD) Cohort
Number analyzed (Participants) | 15 | 12 | 19
months | 4.99 [0.92 to 14.52] | NA [2.66 to NA] — Median and upper CI was not estimable due to insufficient number of events | NA [2.89 to NA] — Median and upper CI was not estimable due to insufficient number of events

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of dosing of study drug up until 30 days after last study dose, up to approximately 10 months.
Description: Assessed in 47 participants who received at least 1 dose of study treatment and were therefore included the Safety Analysis Set.
Arm/Group | Urothelial Cancer (UC) Cohort | Poorly Differentiated Neuroendocrine Carcinomas (PD-NEC) Cohort | Homologous Recombination Deficient-Positive Malignancies Agnostic (HRD) Cohort
All-Cause Mortality (participants affected / at risk) | 9/15 | 3/12 | 5/20
Serious Adverse Events (participants affected / at risk) | 9/15 | 3/12 | 8/20
Other Adverse Events (participants affected / at risk) | 15/15 | 12/12 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Urothelial Cancer (UC) Cohort (N=15) | Poorly Differentiated Neuroendocrine Carcinomas (PD-NEC) Cohort (N=12) | Homologous Recombination Deficient-Positive Malignancies Agnostic (HRD) Cohort (N=20)
Cardiac Arrest (Cardiac disorders) | 0 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 2
Platelet count decreased (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Device occlusion (Product Issues) | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Urothelial Cancer (UC) Cohort (N=15) | Poorly Differentiated Neuroendocrine Carcinomas (PD-NEC) Cohort (N=12) | Homologous Recombination Deficient-Positive Malignancies Agnostic (HRD) Cohort (N=20)
Anaemia (Blood and lymphatic system disorders) | 9 | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 4
Constipation (Gastrointestinal disorders) | 2 | 6 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Eructation (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 6 | 9
Vomiting (Gastrointestinal disorders) | 4 | 2 | 7
Fatigue (General disorders) | 6 | 6 | 8
Localised oedema (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 2
Peripheral swelling (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 2
Abdominal infection (Infections and infestations) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 2 | 2 | 0
Alanine aminotransferase increased (Investigations) | 3 | 4 | 5
Aspartate aminotransferase increased (Investigations) | 3 | 3 | 4
Blood alkaline phosphatase increased (Investigations) | 5 | 4 | 2
Blood bilirubin increased (Investigations) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 3 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 3 | 2 | 2
Gamma-glutamyltransferase increased (Investigations) | 2 | 2 | 1
Lymphocyte count decreased (Investigations) | 4 | 2 | 1
Neutrophil count decreased (Investigations) | 6 | 1 | 3
Neutrophil count increased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 7 | 1 | 6
Procalcitonin increased (Investigations) | 1 | 0 | 0
White blood cell count decreased (Investigations) | 4 | 0 | 2
White blood cell count increased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 5
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 3
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Brain fog (Nervous system disorders) | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 3
Dysarthria (Nervous system disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 2
Dyskinesia (Nervous system disorders) | 1 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 4
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 1 | 1
Incontinence (Renal and urinary disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT05126433/Prot_002.pdf
  • Statistical Analysis Plan (2024-01-19): https://cdn.clinicaltrials.gov/large-docs/33/NCT05126433/SAP_001.pdf